CLINICAL TRIAL: NCT03751176
Title: Phase II Clinical Trial to Evaluate the Efficacy of Second-line FOLFIRI + Panitumumab in Subjects With Wild Type RAS Metastatic Colorectal Cancer Who Have Received FOLFOX + Panitumumab in First-line
Brief Title: Second-line FOLFIRI + Panitumumab in Subjects With Wild Type RAS Metastatic Colorectal
Acronym: BEYOND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Amgen (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-17-01; 2017-004519-38 (EudraCT Number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Clinical trial, phase II; Aged (at least 18 years old); Progression -Free - Survival; Safety; Conversion rate of RAS/BRAF status in liquid biopsy; Chemotherapy regimen; Monoclonal antibody; FOLFIRI; Panitumumab; RAS/BRAF Wild-type
MeSH Terms: interventions — Panitumumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned in a 3:2 ratio to receive FOLFIRI + panitumumab (Group A) or FOLFIRI alone (Group B). Randomization will be stratified by primary tumour location (left vs right).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRI + panitumumab (Experimental): Patients received panitumumab plus FOLFIRI in 14-day cycles until disease progression, unacceptable toxicity, investigator's decision or patient withdrawal of consent, at the following doses:
  * Panitumumab: 6 mg/kg administered by intravenous (IV) infusion over 60 min on days 1 and 14 of every cycle just before administration of chemotherapy
  * FOLFIRI:
  * Irinotecan: 180 mg/m2 as IV infusion over 90 min on day 1
  * Folinic acid: (leucovorin) 200-400 mg/m2 IV over 2 hours on day 1
  * 5-FU: 400 mg/m2 bolus followed by 2400 mg/m2 IV continuous infusion over 46-48 hours on days 1 and 2
  Interventions: Drug: Panitumumab; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-FU
- FOLFIRI (Active Comparator): Patients received FOLFIRI in 14-day cycles until disease progression, unacceptable toxicity, investigator's decision or patient withdrawal of consent, at the following doses:
  * Irinotecan: 180 mg/m2 as IV infusion over 90 min on day 1
  * Folinic acid: (leucovorin) 200-400 mg/m2 IV over 2 hours on day 1
  * 5-FU: 400 mg/m2 bolus followed by 2400 mg/m2 IV continuous infusion over 46-48 hours on days 1 and 2
  Interventions: Drug: Irinotecan; Drug: Folinic acid; Drug: 5-FU

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg will be administered by intravenous (IV) infusion over 60 min on days 1 and 14 of every cycle just before administration of chemotherapy
  Other Names: Vectibix
  Arms: FOLFIRI + panitumumab
Drug: Irinotecan — Irinotecan 180 mg/m2 will be administered as IV infusion over 90 min on day 1
  Other Names: Any marketed
Drug: Folinic acid — Folinic acid 200-400 mg/m2 will be administered as IV infusion over 2 hours on day 1
  Other Names: Any marketed; Leucovorin
Drug: 5-FU — 5-FU will be administered IV 400 mg/m2 bolus followed by 2400 mg/m2 IV continuous infusion over 46-48 hours on days 1 and 2
  Other Names: Any marketed; 5-fluorouracil

SUMMARY:
To estimate progression-free-survival at 6 months in subjects treated in first-line with panitumumab and FOLFOX and with wild type RAS mCRC (metastatic colorectal cancer) confirmed in liquid biopsies before starting second line treatment will be screened for this trial and who have interrupted panitumumab for <3 months (panitumumab continuation). Control arm of subjects treated with FOLFIRI alone will be included.

The combinations of 5-fluorouracil (5-FU) with oxaliplatin (FOLFOX)are considered the backbone chemotherapy for mCRC. Clinical trials have shown the benefit of adding monoclonal antibodies to subjects without mutations in RAS, directed against the epidermal growth factor receptor (EGFR) (cetuximab and panitumumab) to conventional chemotherapy as first-line treatment of mCRC. This trial purposes to study the treatment beyond progression with panitumumab in subjects treated in first-line with an anti-EGFR monoclonal antibody, or rather,the re-introduction of the same targeted therapy after progression to first line.

The clinical hypothesis of this study is that the second-line regimen FOLFIRI + panitumumab, is sufficiently active (defined as a 6-months PFS higher than 30% [based on prior results with second-line FOLFIRI alone] and of at least 50%), justifying further study in this population.

DETAILED DESCRIPTION:
A phase II, multicentre, open-label, randomized two-arm study. Subjects treated in first-line with panitumumab and FOLFOX and with wild type RAS mCRC confirmed in liquid biopsies before starting second line treatment will be screened for this trial. Only subjects who have interrupted panitumumab for < 3 months (panitumumab continuation) will be included.

Eligible subjects will receive FOLFIRI + panitumumab until disease progression, onset of unacceptable drug toxicities, or subject/physician's request to discontinue. A control arm of subjects treated with FOLFIRI alone will be included. Subjects will be assigned in a 3:2 ratio to receive FOLFIRI + panitumumab (Group A) or FOLFIRI alone (Group B). Randomization will be stratified by primary tumour location (left vs right). A blood sample will be obtained at baseline and at disease progression in order to determine the mutational status of RAS/BRAF and other biomarkers.

Tumour response assessment will be performed by the investigator according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria (version 1.1). Subjects will be evaluated for tumour response every 8 weeks until documentation of disease progression. Responding disease will be confirmed no less than 28 days after the criteria for response are first met. Subjects with symptoms suggestive of progressive disease should be evaluated for tumour progression at the time the symptoms occur. After second-line treatment discontinuation, information on subsequent lines of treatments at the physician discretion and survival will be collected in follow-up visits carried out every 12 weeks (± 4 weeks) until the end of the study (approximately 20 months after the inclusion of the last subject in the study).

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman at least 18 years old
2. Capable of understand, sign and date an informed consent approved by an IEC (investigational Ethics Committee)
3. Histologically confirmed adenocarcinoma of the colon or rectum in subjects with metastatic disease
4. Having received a 1st line chemotherapy regimen for mCRC consisting of FOLFOX + panitumumab and having at least achieved stable disease ( i.e., CR (Complete Response) PR (Partial Response) or SD (stable disease) )
5. Wild-type RAS tumour status confirmed in liquid biopsies before starting second-line treatment
6. At least one unidimensionally measurable lesion of at least 10 mm per RECIST criteria (version 1.1)
7. Subjects not candidates for metastasectomy
8. Tumour disease staging according to RECIST (version 1.1) by investigator up to 4 weeks prior to start of study treatment
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
10. Adequate bone marrow function: neutrophils ≥1.5 x109/ L; platelets ≥100 x109/L; haemoglobin ≥9 g/dL
11. Hepatic, renal and metabolic function as follows:

    * Total bilirubin count ≤1.5 x upper limit of normal (ULN), ALT (alanine aminotransferase) and AST (aspartate aminotransferase) <2.5 x ULN; or in case of liver metastasis ALT and AST <5 x ULN
    * Renal function, calculated as creatinine clearance or 24-hour creatinine clearance ≥ 50 mL/min
    * Magnesium > lower limit of normal (LLN) -

Exclusion Criteria:

1. Diagnosis of progressive disease more than 3 months after the last panitumumab administration
2. First-line PFS of less than 3 months
3. Subjects given less than 3 months (consecutive) of first-line panitumumab
4. History of prior or concurrent central nervous system (CNS) metastases
5. History of another primary cancer, except: curatively treated in situ cervical cancer, or curatively resected non-melanoma skin cancer, or other primary solid tumour curatively treated with no known active disease present and no treatment administered for ≥ 5 years before inclusion
6. Prior irinotecan therapy
7. Unresolved toxicities of a previous systemic treatment that, in the opinion of the investigator, cause the subject unfit for inclusion
8. Prior hormonal therapy, immunotherapy or approved or experimental antibody/proteins ≤ 30 days before inclusion (excluding panitumumab)
9. Any investigational agent within 30 days prior to inclusion
10. Evidence of previous acute hypersensitivity reaction, of any grade, to any component of the treatment
11. History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest computerised tomography
12. Acute or subacute intestinal occlusion and/or active inflammatory bowel disease or other bowel disease that causes chronic diarrhoea (defined as grade ≥ 2 diarrhoea according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.03)
13. Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiating study treatment or a history of ventricular arrhythmia
14. History of Gilbert disease or known dihydropyrimidine deficiency syndrome
15. Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
16. Treatment for systemic infection within 14 days before the start of study treatment
17. History of any disease that may increase the risks associated with study participation or may interfere with the interpretation of study results
18. Surgery (excluding diagnostic biopsy or placement of a central venous catheter) and/or radiotherapy within 28 days prior to inclusion in the study.
19. Pregnant or breastfeeding woman
20. Male or female of childbearing age who do not agree with taking adequate contraceptive precautions, i.e. use contraception double barrier (e.g., diaphragm plus condoms) or abstinence during the course of the study and for 6 months after the last administration of study drug for women and 1 month for men
21. The subject is unwilling or unable to meet the requirements of the study
22. Psychological, geographical, familial or sociological conditions that potentially prevent compliance with the study protocol and follow-up schedule. These conditions should be discussed with the subject before inclusion in the trial. -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | 6 months after inclusion
  The proportion of subjects progression free at 6 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 38 months
  Time from randomization to progression or death (Kaplan-Meier estimate)
Overall response rate (ORR) | 38 months
  Proportion of subjects with an objective response (complete or partial response) per RECIST 1.1 criteria
Overall survival (OS) | 38 months
  Time from randomization to the date of death, with participants alive or lost to follow-up at the analysis data cut-off date censored at their last contact date (Kaplan-Meier estimate)
Safety and tolerability. ( assessment will consist of monitoring adverse events (AEs), including serious adverse events (SAEs) and laboratory safety parameters) | 38 months
  Safety assessment will consist of monitoring adverse events (AEs), including serious adverse events (SAEs) and laboratory safety parameters. AEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Biomarkers analysis by liquid biopsies. | 38 months
  Conversion rate of RAS/BRAF status according to liquid biopsy determinations at second-line treatment initiation and at the time of disease progression after second-line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Aparicio, MD, Study Director — Hospital universitari i Politecnic La Fe
Locations (18):
- Spain (18):
  - ICO Girona Dr. Josep Trueta, Girona, Barcelona
  - Hospital de Granollers, Granollers, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital General Universitario de Elche, Alicante, Elche
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - H. Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital de La Ribera de Alzira, Alzira, Valencia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Universtiario la Paz, Madrid
  - CIOCC Sanchinarro, Madrid
  - Complejo Hospitalario de Navarra, Navarro
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GEMCAD (Grupo Español Multidisciplinar en Cancer Digestivo) web page — http://www.gemcad.es/